CLINICAL TRIAL: NCT06467279
Title: Comparison of Patient Outcomes Between Anesthesia Administered Via Target-controlled Infusion Method and Inhalation Anesthesia Method in Pediatric Patients Undergoing Inguinal Hernia Repair
Brief Title: Comparing Inhalation and Total Intravenous Anesthesia Methods
Acronym: TIVA-IHA
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem ÖZ GERGİN, Associate Professor, TC Erciyes University
Other Study IDs: 2022/200; TDK-2022-11979 (Other Grant/Funding Number: TDK-2022-11979)
Record Dates: First submitted 2024-04-16; First posted 2024-06-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Children; Hernia, Inguinal
Keywords: BIS; TIVA; İNFUSİON; İNGUİNAL HERNİA
MeSH Terms: conditions — Hernia, Inguinal | interventions — Anesthetics, Inhalation; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TOTAL INTRAVENOUS ANESTHESIA GROUP: After premedication, anesthesia induction will be performed as per routine. Upon reaching the target Bispectral Index (BIS) level (40-60) and ensuring muscle relaxation, the airway will be secured with an appropriately sized endotracheal tube or laryngeal mask airway (LMA). The target concentration of Propofol in the effect site will be set at 3 mcg/ml using a Target-Controlled Infusion (TCI) device. Controlled ventilation will be conducted with 50% oxygen/air mixture, adjusting mechanical ventilation parameters to maintain End-Tidal Carbon Dioxide (EtCO2) levels between 35-45 mmHg.
  Interventions: Device: Target Controlled İnfusion
- The Patient Group Receiving Inhalation Anesthesia: Patients will be induced with the same anesthesia as Group I, and BIS values will be adjusted to be between 40-60 at the routinely used inhalation gas level of sevoflurane. Patients will be given controlled ventilation with 50% Oxygen/air, and mechanical ventilation materials will be adjusted so that the end tidal carbon dioxide level (EtCO2) will be 35-45 mmHg.
  Interventions: Drug: Inhalation anesthetic

INTERVENTIONS:
Device: Target Controlled İnfusion — TCI (Target-Controlled Infusion) is a method used to maintain the dose and rate of anesthesia drugs within a target concentration range set by the anesthetist. This system delivers drugs intravenously to the patient using a computer-controlled pump. The anesthetist adjusts the drug concentration to achieve the desired depth of anesthesia. This method provides more precise control over anesthesia and facilitates maintaining the depth of anesthesia within the desired range.
  Other Names: TCI
  Groups: TOTAL INTRAVENOUS ANESTHESIA GROUP
Drug: Inhalation anesthetic — In the inhalation anesthesia group, maintenance sevoflurane anesthesia will be applied after routine induction.
  Other Names: Sevoflurane
  Groups: The Patient Group Receiving Inhalation Anesthesia

SUMMARY:
This study compares the effects of anesthesia using target-controlled infusion (TCI) and inhalation methods on pediatric patients undergoing inguinal hernia repair. The main outcomes include intraoperative hemodynamic stability and postoperative recovery characteristics. Sixty children were randomized to receive either total intravenous anesthesia (TIVA) via the Eleveld model or inhalation anesthesia with sevoflurane. The study aims to evaluate which method is safer and more effective in pediatric surgical anesthesia.

DETAILED DESCRIPTION:
This prospective, randomized, controlled study was conducted to evaluate the effects of two anesthesia techniques-target-controlled infusion using total intravenous anesthesia and inhalation anesthesia-on intraoperative hemodynamic stability and postoperative recovery quality in pediatric patients undergoing elective inguinal hernia repair. A total of 60 patients aged 3 to 12 years were randomly assigned to either the TIVA group, which received propofol via TCI using the Eleveld pharmacokinetic model, or the inhalation group, which received sevoflurane-based anesthesia. Standard monitoring included bispectral index (BIS), oxygen saturation (SpO₂), heart rate, and blood pressure measurements. Recovery was assessed using modified Aldrete scoring. A consistent anesthesia depth (BIS 40-60) and standardized ventilatory strategies were maintained for all participants. The aim of this study is to provide comparative data on the safety, efficacy, and recovery profiles of both anesthesia methods in the context of pediatric surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-12 years
* Patients weighing over 10 kilograms
* Patients who will undergo inguinal hernia surgery
* ASA (American Society of Anesthesiologists) classification I and II pediatric patients.

Exclusion Criteria:

* Absence of systemic illness.
* ASA (American Society of Anesthesiologists) classification III pediatric patients.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3-12 with ASA I-II undergoing inguinal hernia repair.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Modified Aldrete Scoring System | after surgery 1 hours
  The effects on recovery were monitored within the first hour of the postoperative period using the Modified Aldrete Scoring System (MASS). Totally 0-10 points can be given by MASS. Higher scores predicts better recovery.

SECONDARY OUTCOMES:
blood pressure (mmHg) | after surgery 1 hours
  The blood pressure of the patients will be measured and recorded in mmHg at five-minute intervals from the beginning until the first postoperative hour.
heart rate (Beats/minute) | after surgery 1 hours
  The heart rate of the patients will be measured and recorded in mmHg at five-minute intervals from the beginning until the first postoperative hour.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem OZ GERGİN, MD, Study Director — TC Erciyes University
Locations (1):
- Özlem OZ GERGİN, Kayseri, Turkey (Türkiye)